CLINICAL TRIAL: NCT04716244
Title: Development of Health Promotion Intervention for Women With Preeclampsia and/or Gestational Diabetes Mellitus
Brief Title: Development of Intervention for Women After Gestational Diabetes or Pre-eclampsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Donna R Zwas, Senior Cardiologist, Hadassah Medical Organization
Other Study IDs: HMO 0858-20
Record Dates: First submitted 2021-01-10; First posted 2021-01-20 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Pre-Eclampsia; Gestational Diabetes
Keywords: Pre-eclampsia; Gestational diabetes; prevention; health promotion; qualitative; intervention-design
MeSH Terms: conditions — Pre-Eclampsia; Diabetes, Gestational | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gestational diabetes: Women who were diagnosed with gestational diabetes within the least year
  Interventions: Other: interview/focus group/questionnaire
- Pre-eclampsia: Women who were diagnosed with pre-eclampsia within the past year
  Interventions: Other: interview/focus group/questionnaire

INTERVENTIONS:
Other: interview/focus group/questionnaire — Prior to the meetings, participants will be asked to fill in a questionnaire with demographic data including age, family status, number of pregnancies, number of children, education, and employment, history of preeclampsia or GDM, family history of CVD, and self-reported height and weight We will conduct up to 8 groups or until we reach saturation of themes. For the teleconference focus groups, the number of participants will be limited to 6 women per group, as recommended from previous research on teleconference focus groups51. The face to face focus groups will include up to -12 women. The expected duration of each group, will last 1-2 hours.
  We will conduct up to 36 in-depth interviews. The expected duration of each interview will last 30 minutes to -1.5 hours.
  Participants will be asked for their consent to record the meetings, audio only. The discussions will be then transcribed. An interview guide will be followed.

SUMMARY:
Our objectives in this qualitative exploratory study:

* To explore the perspectives and preferences of women with preeclampsia and/or GDM history related to a potential health promotion program
* To identify perception of support services post-birth related to health behaviors
* To identify perception of personal and children's risk of future health issues related to GDM and preeclampsia history
* To explore effective intervention strategies and approaches for potential intervention
* To identify barriers and facilitators to adoption and adherence to healthy lifestyles changes in women with preeclampsia and/or GDM history
* Based on our results, literature review and counselling by a panel of health promotion experts, the investigators will design protocol and guidelines for a future interventional health promotion programs

Methods:

Study Design The proposed study consists of a qualitative exploratory study in different populations of women who underwent gestational diabetes or pre-eclampsia.

Health care providers who provide care to women with gestational diabetes and pre-eclampsia will be interviewed to explore effective intervention strategies.

DETAILED DESCRIPTION:
This study aims to explore experiences, views and concerns of women with history of preeclampsia and/or GDM and gain in-depth understanding of the factors that would motivate or deter adoption and adherence to healthy lifestyle and prevention of CVD.

Our objectives in this qualitative exploratory study:

* To explore the perspectives and preferences of women with preeclampsia and/or GDM history related to a potential health promotion program
* To identify perception of support services post-birth related to health behaviors
* To identify perception of personal and children's risk of future health issues related to GDM and preeclampsia history
* To explore effective intervention strategies and approaches for potential intervention
* To identify barriers and facilitators to adoption and adherence to healthy lifestyles changes in women with preeclampsia and/or GDM history
* Based on our results, literature review and counselling by a panel of health promotion experts the investigators will design protocol and guidelines for a future interventional health promotion programs

Methods:

Study Design The proposed study consists of a qualitative exploratory study.

Recruitment

1. Women aged 18-50 years following a pregnancy where they were diagnosed with preeclampsia and/or GDM will participate in this study.
2. Health care providers who provide care to women with gestational diabetes and pre-eclampsia will be interviewed to explore effective intervention strategies.

Recruitment site 1: the investigators will conduct focus groups in Hebrew and Arabic with women after preeclampsia and/or GDM who gave birth in the Hadassah medical center or are participating in the Hadassah postpartum clinic for patients with complicated pregnancies. Separate focus groups will be conducted for women with prior preeclampsia and for women with GDM history.

The eligible women will be approached by the study investigator and will be informed about the study. The interested women will be recruited to participate in this study and will be asked to sign a consent form.

Those not able to participate in focus groups will be invited to share their experience through in-depth interviews.

Given the restrictions imposed by the Covid-19 pandemic, as well as the evidence about the difficulty among post-partum women to attend face-to-face interviews50, participants will be offered to participate in either on-site, face to face interviews in Hadassah or teleconference-based interviews (by phone or secured online meeting forms such as zoom meetings).

The investigators will ensure that the face to face groups/ interviews will be conducted in accordance with the physical-distancing instructions of the ministry of health due to Covid-19 pandemic.

The women will be contacted by the research team within 1 year from discharge. The investigators will contact them through the phone or e-mail to plan their participation in the focus groups/ in depth interviews. The interviews will take place within 12 months from the discharge.

Recruitment site 2: the investigators will recruit ultra-Orthodox (Haredi) and Arab participants through community centers from different neighborhoods in Jerusalem.

Invitation to participate in the interviews will be published using posters and/or direct contact with the women by the community-center's staff. The investigators will recruit women that participate in post-partum mothers' programs through community centers, in the Haredi and Arab neighborhoods. The eligible and interested women will be recruited to participate in the study and will be asked to sign a consent form prior to the interview. The women will sign consent before the meetings or phone consent for teleconference/ phone meetings.

Inclusion criteria/ Exclusion criteria

The investigators will recruit women:

* Who gave birth in Hadassah medical center, Jerusalem (within 12 months of a live birth) or participating to the Hadassah postpartum clinic for patients with complicated pregnancies
* After a pregnancy where women were diagnosed with preeclampsia and/or GDM (diagnosed) within 12 months post-partum
* Between 18 and 50 years old
* That will be able to communicate in Hebrew or Arabic

In the community centers, the investigators will recruit women:

* After a pregnancy where women were diagnosed with preeclampsia and/or GDM (diagnosed) within 12 months of a live birth
* Between 18 and 50 years old
* That will be able to communicate in Hebrew or Arabic The investigators will exclude women with serious complications of preeclampsia and or/GDM as perinatal mortality or multi-organ failure.

The investigators will interview health care practitioners who provided health care within the Hadassah system and outside clinics.

Quantitative component:

Prior to the meetings, participants will be asked to fill in a questionnaire (will take approximately 10 minutes) . The questionnaire consists on the following sections:

Demographic data including age, family status, number of pregnancies, number of children, education, and employment History of disease: preeclampsia or GDM, family history of CVD Self -reported height and weight

Participants, who will be interviewed through tele-conference, will receive the questionnaire through electronically and will be asked to fill it prior to the interview. The questionnaire will be filled out using a participant ID which is de-identified, and will be collected through the Nemala system which is encrypted and secure according to Ministry of Health and Helsinki committee recommendations. Participants who will be unable to fill in electronically (Haredi population) will complete the questionnaire by phone. For on-site and face to face interviews, participants will be administered a print copy or the online questionnaire using a computer or tablet, using the de-identified participant identification, and will be asked to fill it prior to the interview.

Number of participants - up to 100 Focus group discussions: the investigators will conduct up to 8 groups or until the investigators reach saturation of themes. For the teleconference focus groups, the number of participants will be limited to 6 women per group, as recommended from previous research on teleconference focus groups51. The face to face focus groups will include up to -12 women. The expected duration of each group, will last 1-2 hours.

In-depth interviews: The investigators will conduct up to 36 in-depth interviews. The expected duration of each interview will last 30 minutes to -1.5 hours.

The investigators will recruit up to 100 women in total for focus groups and in-depth interviews. Each participant will be interviewed only once, in a focus group or in-depth interview, depending on her preference.

Prior to the interviews, the interviewer will explain again the purpose of the study. Interviews will be conducted by researchers from the Linda Joy Pollin center who have a previous experience conducting qualitative studies.

Participants will be asked for their consent to record the meetings, audio only. The discussions will be then transcribed without any identification information of the participants and the recordings will be destroyed afterwards. An interview guide was prepared by the research staff (see attached the interview guides- for focus groups and in-depth interviews).

To maintain confidentiality, the investigators will use first names only during the face to face/ online meeting forms -zoom meetings.

Data analysis

Focus groups and in-depth interviews will be recorded, transcribed and analyzed by investigator according to a thematic analysis:

1. Total impression - from chaos to themes
2. Identifying and sorting meanings units - from themes to codes
3. Condensation - from code to meaning
4. Synthesizing - from condensation to descriptions and concepts

Data Storage In order to maintain confidentiality, all paper data will be stored in a double locked storage space at Hadassah hospital. No identifying information will be collected on the data itself (either electronic or paper), aside from a coding number. Any documentation of focus groups/ in-depth interviews outcomes will not include identifying information.

ELIGIBILITY:
Inclusion Criteria:

* women:

  * within 12 months of a live birth
  * After a pregnancy where women were diagnosed with preeclampsia and/or GDM (diagnosed) within 12 months post-partum
  * Between 18 and 50 years old

Exclusion Criteria:

- We will exclude women with serious complications of preeclampsia and or/GDM as perinatal mortality or multi-organ failure.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients who identify as female and who have given birth.
Study Population: Women within 12 months of gestational diabetes or pre-eclampsia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Identification of four consistent themes on thematic qualitative analysis | 12 months
  Themes are general propositions that emerge from diverse and detail-rich experiences of participants and provide recurrent and unifying ideas regarding the subject of inquiry. Themes evolve from the conceptual codes and subcodes as in the case of taxonomy and also from the relationship codes, which tag data that link concepts to each other.

CONTACTS AND LOCATIONS:
Overall Officials: Donna Zwas, MD MPH, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Please Select An Option Below, Israel

IPD SHARING:
Plan to Share IPD: No
Given the confidential nature of personal interviews, the de-identified thematic analysis will be made available on request of investigators with active GCP